CLINICAL TRIAL: NCT07176312
Title: - ZANGEA - Phase II Study of Zanidatamab in Combination With Pembrolizumab and Chemotherapy in HER2 and PD-L1 Positive Metastatic Gastroesophageal Adenocarcinoma (GEA) Patients
Brief Title: Zanidatamab in Combination With Pembrolizumab and Chemotherapy in HER2 and PD-L1 Positive Metastatic Gastroesophageal Adenocarcinoma (GEA) Patients
Acronym: ZANGEA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKF/AIO-ZANGEA; 2025-522718-22-00 (EU CTIS Number); AIO-STO-0425/ass (Other: AIO Arbeitsgemeinschaft Internistische Onkologie in der Deutschen Krebsgesellschaft e.V.); IKF090 (Other: Frankfurter Institut für Klinische Krebsforschung IKF GmbH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Gastroesophageal Adenocarcinoma; First Line Therapy; HER2 + Gastric Cancer; PDL-1; Metastases
Keywords: GEA; Gastroesophageal adenocarcinoma; first line therapy; HER2-positive; PD-L1 positive
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — zanidatamab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, open-label, multicenter, multinational phase II study. All patients receive zanidatamab in combination with pembrolizumab and mFOLFOX.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanidatamab plus pembrolizumab and mFOLFOX (Experimental): Single Arm with Zanidatamab Q2W in combination with pembrolizumab Q6W and mFOLFOX Q2W
  Interventions: Drug: Zanidatamab; Drug: Pembrolizumab; Drug: mFOLFOX

INTERVENTIONS:
Drug: Zanidatamab — Zanidatamab 1,200 mg (patients <70 kg at baseline) or 1,600 mg (patients ≥70 kg at baseline), administered i.v. on day 1 of each 2-week cycle (Q2W)
Drug: Pembrolizumab — Pembrolizumab 400 mg, administered i.v. on day 1 of every third cycle (Q6W)
Drug: mFOLFOX — modified FOLFOX with Oxaliplatin 85 mg/m2 i.v. on day 1; Folinic Acid 400 mg/m2 i.v. on day 1; 5-FU 2,400 mg/m2 i.v. continuous infusion over 48 hours (no bolus!) on days 1 and 2 of each 2-week cycle (Q2W)

SUMMARY:
The ZANGEA trial is a open-label, single arm, multicenter phase II trial assessing the efficacy of zanidatamab in combination with pembrolizumab and chemotherapy in patients with metastatic gastroesophageal adenocarcinoma (GEA). The patients need to be previously untreated in the palliative setting and tested positive for HER2 and PD-L1.

DETAILED DESCRIPTION:
The ZANGEA trial is designed as a single arm phase II study, which aims to estimate the therapeutic efficacy of the experimental regimen zanidatamab in combination with pembrolizumab and chemotherapy in HER2 and PD-L1 positive metastatic gastroesophageal adenocarcinoma (GEA) without previous palliative treatment.The primary objective is to evaluate the efficacy of this treatment, secondary objectives are to further determine the efficacy, to evaluate safety and tolerability and to assess quality of life (QoL).

In addition, two explorative objectives are defined: preplanned matched-pair analyses comparing the study arm to a historical study arm with trastuzumab, chemotherapy and PD-1 inhibitor (AIO INTEGA) in terms of efficacy, tolerability, and translational data and to correlate analysis between selected molecular tumor, serum and microbiome parameters and clinical data to identify molecular biomarkers predictive for tumor response, toxicity, and survival.

A total of 80 patients will be enrolled in approx. 30 study sites in Germany and Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patient* has signed and dated a written informed consent form in accordance with regulatory and institutional guidelines and approved by an institutional Review Board / Independent Ethics Committee. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
* Patient is, in the investigator's judgement, willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Patient is ≥ 18 years of age at time of signing the written informed consent.
* Patient has been diagnosed with histologically confirmed unresectable advanced/metastatic HER2-positive (defined as IHC 3+ or IHC 2+ with ISH+) and PD-L1-positive (combined positive score CPS ≥ 1) gastroesophageal adenocarcinoma per local standard assessment of new or archival tumor tissue. Results of local HER2 and PD-L1 assessment will be retrospectively confirmed by central pathological re-assessment.

Note: In case of metachronous metastases, particularly in case of prior treatment with PD-(L)1-antibodies, a fresh re-biopsy should be performed for immunohistochemistry testing (local pathology), if feasible.

* Patient has assessable disease (measurable or non-measurable) per RECIST v1.1.
* Patient did not receive previous palliative treatment. Prior adjuvant or neoadjuvant chemotherapy, immunotherapy, radiotherapy and/or chemoradiotherapy (but not anti HER2-targeted treatment) are permitted as long as the last administration of the last regimen (whichever was given last) occurred at least 6 months prior to enrolment.
* Patient has ECOG performance status ≤ 1.
* Patient has adequate hepatic, renal and hematologic functions:

  1. Absolute number of neutrophils (ANC) ≥ 1.5 x 10^9/L
  2. Platelets ≥ 100x10^3/µL
  3. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (measured by 24 h urine) ≥ 30 mL/min (i.e., if serum creatinine level is > 1.5 x upper limit of normal (ULN), then a 24-hour urine test must be performed to check the creatinine clearance to be determined.
  4. AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN (or ≤ 5.0 x ULN if liver metastases are present)
  5. Total Bilirubin ≤ 1.5 x ULN (or < 3.0 x ULN in case of prior liver involvement or Gilbert's Syndrome)
* Patient has adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotrophin [hCG]) within 7 days prior to the start of study drug. Women must not be breastfeeding. WOCBP must use a highly effective method(s) of contraception during the treatment period and for 4 months after last dose of zanidatamab and/or pembrolizumab, or 6 months after the last dose of chemotherapy, whichever occurs last. Males who are sexually active with WOCBP must agree to remain abstinent or follow instructions for method(s) of contraception during the treatment and for 4 months after the last dose of zanidatamab and/or pembrolizumab, or 6 months after the last dose of chemotherapy, whichever occurs last. In addition, male subjects must be willing to refrain from sperm donation during this time.

  * There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.

Exclusion Criteria:

* Patient has any known contraindication including allergy or hypersensitivity to the trial drugs or any constituent of the products as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies.
* Patient received prior anti HER2-targeted treatment for GEA.
* Patient has malignancies other than the disease under study within 5 years prior to inclusion, except for those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
* Patient has untreated known CNS metastases. Patient is eligible, if previous CNS metastases are adequately treated and patient has neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for ≥ 2 weeks prior to enrolment, and did not receive corticosteroids, or is on a stable or decreasing dose of < 10 mg daily prednisone (or equivalent) for ≥ 2 weeks prior to inclusion.
* Patient has abnormal baseline left ventricular ejection fraction (LVEF < 50 %), assessed by echocardiogram, multigated acquisition (MUGA) scan, or cardiac magnetic resonance imaging (MRI) scan.
* Patient has active, known, or suspected autoimmune disease. Exception: Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the medical expert/sponsor be consulted prior to signing informed consent.
* Patient has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of trial drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patient has persisting toxicity related to prior therapy (NCI CTCAE v.5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Patient has any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with trial participation, trial drug administration, or would impair the ability of the patient to receive trial drug.
* Patient has significant acute or chronic infections including, among others:
* Any positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Patient has history of allogeneic tissue / solid organ transplant.
* Patient has been incarcerated or involuntarily institutionalized by court order or by the authorities [§ 40 Abs. 1 S. 3 Nr. 4 AMG].
* Patient is unable to consent because he/she does not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
* Patient has evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the trial medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of trial results.
* Patient currently participates in any other interventional clinical study within 30 days before the first administration of the investigational product or at any time during the trial, unless it is an observational (non-interventional) study, or during the follow-up period of an interventional study with last dose of investigational product ≥28 days prior to enrolment in this trial.
* Patient has a known complete absence of dihydropyrimidine dehydrogenase (DPD) activity or use of any medications known to inhibit DPD (including brivudine, sorivudine and analogs) within 4 weeks prior to enrolment.
* Female patients, who are pregnant or breast feeding or planning to become pregnant within and 6 months after the end of treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of zanidatamab in combination with pembrolizumab and chemotherapy in previously untreated HER2 and PD-L1 positive metastatic gastroesophageal adenocarcinoma (GEA) | 12 months after start of trial medication
  Progression-free survival rate at 12 months (PFS@12), estimated using Kaplan Meier method and defined as proportion of patients alive and progression-free 12 months after start of trial medication

SECONDARY OUTCOMES:
To further determine the efficacy of zanidatamab in combination with pembrolizumab and chemotherapy in metastatic GEA. | up to 42 months after enrolment
  Overall response rate (ORR), defined as proportion of patients achieving complete or partial response (CR/PR) acc. to RECIST v1.1.
  Disease control rate (DCR), defined as proportion of patients achieving CR, PR, or stable disease (SD) acc. to RECIST v1.1.
  Duration of response (DoR), defined as time from response initiation (when either CR or PR is first determined) to disease progression acc. to RECIST v1.1 or death due to any cause.
  Progression-free survival (PFS), defined as time from first treatment until date of progression acc. to RECIST v1.1 or death due to any cause.
  Overall survival (OS), defined as time from first treatment until date of death due to any cause.
To evaluate safety and tolerability of zanidatamab in combination with pembrolizumab and chemotherapy in metastatic GEA. | up to 25 months after first study treatment
  Assessment of safety of the treatment as determined by the incidence, nature, causality, frequency, timing, and severity of adverse events using NCI CTCAE v5.0
Assessment of quality of life (QoL) data | up to 42 months after first study treatment
  Assessment of QoL during treatment and follow-up using EORTC QLQ-C30 and EQ-5D-5L questionnaires.

OTHER OUTCOMES:
Preplanned matched-pair analyses comparing the study arm to a historical study arm | after end of study of all patients, up to 54 months after first patient enrolment
  Preplanned matched-pair analyses comparing the study arm to a historical study arm with trastuzumab, chemotherapy and PD-1 inhibitor (AIO INTEGA) in terms of efficacy, tolerability, and translational data
correlation analysis between selected molecular tumor, serum and microbiome parameters and clinical data to identify molecular biomarkers predictive for tumor response, toxicity, and survival. | after end of study of all patients, up to 54 months after first patient enrolment
  To correlate analysis between selected molecular tumor (such as CPS cut-offs ≤ 5 and >5 - 10, as well as HER2 IHC2+/ISH+ vs. IHC3+), serum and microbiome parameters and clinical data to identify molecular biomarkers predictive for tumor response, toxicity, and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH; Alexander Stein, Prof. Dr., Principal Investigator — Hämatologisch-Onkologische Praxis Eppendorf University Cancer Center Hamburg
Locations (20):
- Germany (20):
  - Charité CVK, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Städtisches Klinikum Dresden, Dresden
  - Evang. Kliniken Essen Mitte, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Göttingen, Göttingen
  - Hämatologisch Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - St. Anna Hospital Herne, Herne
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin Mainz, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum rechts der Isar der TU München, München
  - LMU Klinikum München Großhadern, München
  - MVZ für Hämatologie und Onkologie Ravensburg, Ravensburg
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No